CLINICAL TRIAL: NCT05833295
Title: Electrophysiological and Clinical Effects of Walking Downhill in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAR.FTR.ST
Record Dates: First submitted 2023-03-28; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Patients will be randomized into 3 groups. Clinical and electrophysiological tests before and after walking sessions will be performed by an unannounced researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Walking on flat ground (Experimental): Patients will walk for 20 minutes at a 0% slope.
  Interventions: Procedure: Walking on flat ground
- -%7.5 Downhill walking (Experimental): They will walk downhill for 20 minutes at a -(negative)7.5% gradient.
  Interventions: Procedure: Downhill walking
- -%15 Downhill walking (Experimental): They will walk downhill for 20 minutes at a -(negative)15% gradient.
  Interventions: Procedure: Downhill walking

INTERVENTIONS:
Procedure: Downhill walking — Change in the H/M ratio after a downhill walk.
  Arms: -%15 Downhill walking; -%7.5 Downhill walking
Procedure: Walking on flat ground — Change in the H/M ratio after a Walking on flat ground
  Arms: Walking on flat ground

SUMMARY:
investigation of the effects of walking for 20 minutes on the acute H/M ratio on flat ground, downhill slopes at -7.5 degrees and -15 degrees in patients who have had a stroke, have spasticity and are ambulatory.

At the same time, the aim of the study is to obtain the clinical effectiveness of this walking pattern and control of the H/M ratio by checking the H/M ratio again after 5 sessions and 20 minutes of walking for the patients participating in the study.

DETAILED DESCRIPTION:
Participants will wear a seat belt connected to an overhead support and will walk on a treadmill with a dual-band instrument at a sampling frequency of 2000 Hz. The seat belt will only serve as a safety mechanism in case of a fall and will not support any body weight while walking. Each participant will walk for 20 minutes under one of 3 slope conditions; treadmill walking on 0° flat ground, , downhill walking with treadmill on -7.5° slope and downhill walking with treadmill on -15° slope.

First, by asking the participants to walk at their comfortable speed for straight walking on the treadmill with tools, the walking speed will be determined and carried out at the specified speeds. All self-selected walking speeds will be determined in two 30-second trials. During the 20-minute walk for each condition, if the participant needs to slow down, the speed of the treadmill will be reduced to adapt to this, and the average walking speed during the 20-minute walking session will be reported. Pulse and blood pressure will be monitored before, during and after the walk.

All participants will be evaluated with modified asworth scale, modified tardeu scale, 2 minute walking test, modified rankin scale, timed get up and walk test, fatigue impact scale, stroke impact scale, berg balance scale, fugl meyer assessment scale before treatment.

Patients will be randomized into 3 groups. Then, the H / M ratio will be looked at in all 3 groups. After the first walking session, the H / M ratio will be repeated. after completing the 5-session walking program, clinical and electrophysiological tests will be repeated.

ELIGIBILITY:
Inclusion Criteria:

patients diagnosed with stroke between the ages of 18 and 65 Dec

Exclusion Criteria:

* Other neurological disorders,

  * Expressive or receptive aphasias,
  * Severe heart disease,
  * A history of poorly controlled diabetes,
  * Active cancer,
* Those who have been injected with botilinum toxin in the last 3 months,

  * Orthopedic conditions affecting the legs, a history of hip or knee replacement,
  * Serious simultaneous medical problems, such as peripheral nerve damage
* Inability to comprehend verbal instructions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-04-24 (Estimated); Primary Completion 2023-05-24 (Estimated); Study Completion 2024-04-24 (Estimated)

PRIMARY OUTCOMES:
the change in the H/M ratio after a 20-minute walk. | Day 0: Before the walk
  Each participant will be evaluated for changes in the H/M ratio with an EMG device before the walk, on the 1st day of the walk, and on the 5th day of the walk.
the change in the H/M ratio after a 20-minute walk. | Day 1: First day of 20-minute walk
  Each participant will be evaluated for changes in the H/M ratio with an EMG device before the walk, on the 1st day of the walk, and on the 5th day of the walk.
the change in the H/M ratio after a 20-minute walk. | Day 5: The fifth day of the 20-minute walk
  Each participant will be evaluated for changes in the H/M ratio with an EMG device before the walk, on the 1st day of the walk, and on the 5th day of the walk.

SECONDARY OUTCOMES:
Modified Asworth Scale | Day 0: Before the walk
  Modified Asworth Scale is a spasticity assessment test. It contains 4 points in total. As the score increases, the degree of spasticity increases.
Modified Asworth Scale | Day 5: The fifth day of the 20-minute walk
  Modified Asworth Scale is a spasticity assessment test. It contains 4 points in total. As the score increases, the degree of spasticity increases.
Modified Tardeu Scale | Day 0: Before the walk
  Modified Tardeu Scale is a spasticity assessment test. It contains 5 points in total. As the score increases, the degree of spasticity increases.
Modified Tardeu Scale | Day 5: The fifth day of the 20-minute walk
  Modified Tardeu Scale is a spasticity assessment test. It contains 5 points in total. As the score increases, the degree of spasticity increases.
Walking test | Day 0: Before the walk
  2 minute walking test
Walking test | Day 5: The fifth day of the 20-minute walk
  2 minute walking test
Walking capacity | Day 0: Before the walk
  Timed Get Up and Walk Test
Walking capacity | Day 5: The fifth day of the 20-minute walk
  Timed Get Up and Walk Test
The Fatigue Effect Scale | Day 0: Before the walk
  The fatigue effect scale consists of 9 questions. Each question gets points between 0 and 7. The total score is divided by the number of questions. If the result is greater than 6.1, it is defined as chronic fatigue.
Fatigue | Day 5: The fifth day of the 20-minute walk
  The fatigue effect scale consists of 9 questions. Each question gets points between 0 and 7. The total score is divided by the number of questions. If the result is greater than 6.1, it is defined as chronic fatigue.
Stroke impact scale | Day 0: Before the walk
  Stroke Impact Scale; patients' quality of life after stroke to assess their perception by themselves or their caregivers This scale consists of 8 subsections and 59 questions. each one question is a 5-point Likert scale of difficulty experienced in the past week.
  It is scored by evaluation on the scale. each section The score ranges from 0 to 100. In addition, the stroke impact scale has 8 subsections.
  0-100 point visual analog of the perception of recovery after stroke. scale (0: No improvement, 100: Full recovery)
Stroke impact scale | Day 5: The fifth day of the 20-minute walk
  Stroke Impact Scale; patients' quality of life after stroke to assess their perception by themselves or their caregivers This scale consists of 8 subsections and 59 questions. each one question is a 5-point Likert scale of difficulty experienced in the past week.
  It is scored by evaluation on the scale. each section The score ranges from 0 to 100. In addition, the stroke impact scale has 8 subsections.
  0-100 point visual analog of the perception of recovery after stroke. scale (0: No improvement, 100: Full recovery)
Berg Equilibrium Scale | Day 0: Before the walk
  It is a scale that includes 14 instructions and is scored between 0-4 by observing the patient's performance for each instruction. While 0 points are given when the patient cannot do the activity at all, 4 points are given when the patient completes the activity independently. The highest score is 56, with 0-20 points indicating balance disorder, 21 40 points indicating an acceptable balance, 41-56 points indicating a good balance. It takes between 10 and 20 minutes to complete the scale.
  It is a scale that includes 14 instructions and is scored between 0-4 by observing the patient's performance for each instruction. While 0 points are given when the patient cannot do the activity at all, 4 points are given when the patient completes the activity independently. The highest score is 56, with 0-20 points indicating balance disorder, 21 40 points indicating an acceptable balance, 41-56 points indicating a good balance. It takes between 10 and 20 minutes to complete the scale.
Berg Equilibrium Scale | Day 5: The fifth day of the 20-minute walk
  It is a scale that includes 14 instructions and is scored between 0-4 by observing the patient's performance for each instruction. While 0 points are given when the patient cannot do the activity at all, 4 points are given when the patient completes the activity independently. The highest score is 56, with 0-20 points indicating balance disorder, 21 40 points indicating an acceptable balance, 41-56 points indicating a good balance. It takes between 10 and 20 minutes to complete the scale.
Fugl-Meyer Assessment Scale | Day 0: Before the walk
  The full version of FMRS assesses five domains: motor function, balance, sensory function, range of motion (ROM) and joint pain. In the full version of the scale, when all subscales (sensory function 24 points, balance 14 points, ROM 44 points, joint pain 44 points and motor-coordination 100 points) are added, the maximum total score is 226. The motor-coordination subscale is a maximum of 66 points for the upper extremity and a maximum of 34 points for the lower extremities. Higher scores indicate better motor recovery. Each item is scored with a 3-point ordinal scale (0: unable at all, 1: partially able, 2: fully able). When items related to coordination and speed are not included in the evaluation in the lower extremity motor-coordination subscale, it is specified as the lower extremity motor subscale and its maximum score is evaluated out of 28.
Fugl-Meyer Assessment Scale | Day 5: The fifth day of the 20-minute walk
  The full version of FMRS assesses five domains: motor function, balance, sensory function, range of motion (ROM) and joint pain. In the full version of the scale, when all subscales (sensory function 24 points, balance 14 points, ROM 44 points, joint pain 44 points and motor-coordination 100 points) are added, the maximum total score is 226. The motor-coordination subscale is a maximum of 66 points for the upper extremity and a maximum of 34 points for the lower extremities. Higher scores indicate better motor recovery. Each item is scored with a 3-point ordinal scale (0: unable at all, 1: partially able, 2: fully able). When items related to coordination and speed are not included in the evaluation in the lower extremity motor-coordination subscale, it is specified as the lower extremity motor subscale and its maximum score is evaluated out of 28.

CONTACTS AND LOCATIONS:
Locations (1):
- Mamara Üniversitesi Tıp Fakültesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No